CLINICAL TRIAL: NCT06038981
Title: Assessment of the Impact of Perioperative Administration of Tranexamic Acid on Bleeding After Sleeve Gastrectomy - a Randomized Clinical Trial
Brief Title: Assessment of the Impact of Perioperative Administration of Tranexamic Acid on Bleeding After Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TXA_SG
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hemorrhage, Surgical; Bariatric Surgery; Tranexamic Acid
Keywords: bariatric surgery; Hemorrhage; Tranexamic Acid
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG). (No Intervention): no tranexamic acid administration.
- TXA group. (Experimental): Administration of 1g tranexamic acid intravenous bolus, after anesthesia was introduced.
  Interventions: Drug: Administration of 1g tranexamic acid intravenous bolus, after anesthesia was introduced

INTERVENTIONS:
Drug: Administration of 1g tranexamic acid intravenous bolus, after anesthesia was introduced — The systemic use of tranexamic acid (TXA) has been shown to be effective in many types of surgery, reducing the incidence of post-operative bleeding and thereby reducing the rate of reoperation.
  To evaluate if TXA systemic administration reduces postoperative blood loss in bariatric surgeries (sleeve gastrectomy operation)
  Arms: TXA group.

SUMMARY:
Enhanced recovery after bariatric surgery imposes a significant reduction in length of hospital stay. However beneficial for the overall recovery it reduces the hospital observation time. after a laparoscopic surgery during which one of the longest resection line in surgery or anastomosis are created. Therefore, discovering possible safe and effective ways of pharmacologically reducing surgical blood loss and reducing the risk of postoperative bleeding would be an invaluable addition to the protocol. The systemic use of tranexamic acid (TXA) has been shown to be effective in many types of surgery, reducing the incidence of post-operative bleeding and thereby reducing the rate of reoperation.

DETAILED DESCRIPTION:
Aim:

To evaluate if TXA systemic administration reduces postoperative blood loss in bariatric surgeriessleeve gastrectomy operation.

Material and methods:

A single-blind randomized clinical trial in the high-volume bariatric center of excellence.

Patients undergoing highly standardized bariatric procedures, meeting the inclusion and exclusion criteria were included in the study, sample size determined by power study evaluation.

Randomization scheme was a weekly surgery schedule. Patients were randomized to 2 groups: TXA (administration of 1g tranexamic acid intravenous bolus, after anesthesia was introduced) od CG (no tranexamic acid administration).

Patients were evaluated on the postoperative day 1 by standard lab tests included in the center's protocol, additionally measuring the volume of drainage and heamoglobin concentration in the drainage sample.

1-month follow-up observation involving interviewing, examining and conducting lab tests of the study group was provided to determine the safety profile and possible occurrence of TXA complications.

ELIGIBILITY:
Inclusion Criteria:

* Participant were adults qualified for bariatric procedure

Exclusion Criteria:

* Primary (pre-operative) exclusion criteria were as follows:
* Usage of anticoagulative agents in the perioperative period including:
* Indirect thrombin inhibitors (Fondaparinux, UFH, LMWH in therapeutic dosing)
* Direct inhibitors of factor Xa (NOAC)
* Direct thrombin inhibitors (Dabigatran)
* Vitamin K Antagonists (VKA: acenokumarol, warfarin)
* Platelet aggregation inhibitors (excluding ASA in dosing 75mg per day)
* P2Y12 receptor inhibitors
* Prior diagnosis of congenital or acquired blood coagulation disorders
* Diagnosed allergic reactions to TXA in medical history
* Chronic Kidney Disease in stage G3 or higher
* Chronic hemodialysis
* Haematuria in medical history
* Seizures in medical history

To achieve the most homogenous group of patients and to reduce possible bias due to additional interventions occurring during the operation - further, postoperative exclusion criteria were introduced:

Performed operation other than laparoscopic sleeve gastrectomy (LSG) Necessity of TXA administration in the postoperative period Additional, supplementary heamostatic materials and methods were used during the operation - deviation from the standard operation protocol such as: use of oxidized regenerative cellulose (ORC), cyanoacrylate laparoscopic bioglue (IfabondÒ, Peters Surgical), staple-line reinforcement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Blood loss. | First postoperative day.
  Patients were evaluated on the postoperative day 1 by standard lab tests included in the center's protocol, additionally measuring the volume of drainage and heamoglobin concentration in the drainage sample.

SECONDARY OUTCOMES:
TXA complications. | One month.
  1-month follow-up observation involving interviewing, examining and conducting lab tests of the study group was provided to determine the safety profile and possible occurrence of TXA complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol and SAP will be available soon online.